CLINICAL TRIAL: NCT00795314
Title: Propofol-butorphanol Combined Anesthesia During Uterine Curettage on Abortion
Brief Title: Propofol-butorphanol Anesthesia During Uterine Curettage
Acronym: PABADUC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-2008-FY10MZ31; NJFY0811-MZ02
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Abortion; Curettage
Keywords: Opioids; General anesthesia
MeSH Terms: interventions — Fentanyl; Butorphanol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Propofol-fentanyl combined anesthesia
  Interventions: Drug: Fentanyl Citrate
- 2 (Experimental): Propofol-butorphanol combined anesthesia
  Interventions: Drug: Butorphanol Tartrate

INTERVENTIONS:
Drug: Fentanyl Citrate — Combined anesthesia with propofol (2-2.5mg/kg) and fentanyl (5 μg)
  Other Names: Actiq®; Fentora TM; Duragesic®
  Arms: 1
Drug: Butorphanol Tartrate — Combined anesthesia with propofol (2-2.5 mg/kg) and butorphanol (1mg)
  Other Names: Torbugesic®; Torbutrol®
  Arms: 2

SUMMARY:
Uterine curettage is usually performed under the anesthesia of propofol-fentanyl or para-cervical block,of which generally has significant incidence of respiratory depression which increases the demand on intraoperative monitoring, or has unavoidable insufficient blockade which results in intraoperative suffering of pain. Butorphanol is an analgesic with combined effects on mu and kappa opioid receptors leading to a role as analgesia and sedation. The investigators hypothesized that combined propofol with butorphanol during uterine curettage would produce optimal effectiveness of these two drugs by adding sedative and analgesic effects together. In addition, it would decrease the intraoperative consumption of propofol without increase the incidence of side effects. Furthermore, such combination would alleviate postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* ASA status I-II;
* Performing abortion operation (medical- or drug-induced);
* Requiring painless abortion;

Exclusion Criteria:

* < 19yrs, and >= 45yrs;
* History of central active drugs administration;
* Drug abuse;
* Hypertension;
* Diabetes;
* Any other chronic diseases;
* Allergy to the study drugs;
* Habit of over-volume alcohol drinking;
* Records of history of centrally active drug use and psychiatry;
* Any organic disorders.

Ages: 19 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2008-11; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Intraoperative awareness | During the whole process of anesthesia

SECONDARY OUTCOMES:
Bispectral Index (BIS) value | During the whole process of anesthesia
Anesthetic consumptions | From the start of operation to the end of surgical procedures
Postoperative pain | Since the end of the operation to 48 h follow-up.
Postoperative bleeding | Since the end of operation to 48 h follow-up

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Chair — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China